CLINICAL TRIAL: NCT04188249
Title: A Prospective Multicenter Registry of Golimumab in Chinese Patients With Rheumatoid Arthritis
Brief Title: Effectiveness and Adherence of Golimumab in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CNTO148ARA4012
Record Dates: First submitted 2019-06-27; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-06

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RA patients: Patients (or a representative) must provide informed consent before any procedures occur.
  1. Main Inclusion Criteria:
     * 18 years and older
     * Fulfil the ACR/EULAR classification criteria for RA in 2010
     * Patients able to understand and complete self-evaluation questionnaires.
  2. General Exclusion Criteria:
     * Contraindications for golimumab
     * Prior exposure to TNFi/JAKi
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — This multicenter (12 centers), prospective program will register 200 RA patients routinely receiving golimumab treatment. Doctor will record the disease evaluation, concomitant drug, adverse events and laboratory tests based on patient's visit till they withdraw from clinical visit. Doctor will still collect above information whether patient interrupt or stop golimumab till the end of program or patient withdraw permanently.

SUMMARY:
This will be a prospective, observational, single-arm, registry study based on data received from Chinese Registry of rheumatoid arthritis (CREDIT) database to register 200 Chinese RA patients treated with golimumab in one year. Patient characteristic, clinical effectiveness and drug adherence of golimumab will be evaluated.

DETAILED DESCRIPTION:
This multicenter (12 centers), prospective program will register 200 RA patients routinely receiving golimumab treatment. Doctor will record the disease evaluation, concomitant drug, adverse events and laboratory tests based on patient's visit till they withdraw from clinical visit. Doctor will still collect above information whether patient interrupt or stop golimumab till the end of program or patient withdraw permanently.

ELIGIBILITY:
Inclusion Criteria:

* - 18 years and older
* Fulfil the ACR/EULAR classification criteria for RA in 2010
* Patients able to understand and complete self-evaluation questionnaires.

Exclusion Criteria:

* - Contraindications for golimumab
* Prior exposure to TNFi/JAKi

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter (12 centers), prospective program will register 200 RA patients routinely receiving golimumab treatment. Doctor will record the disease evaluation, concomitant drug, adverse events and laboratory tests based on patient's visit till they withdraw from clinical visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of low disease activity (CDAI) at week 12 | At week 12
  Low disease activity is defined as crohn's disease activity index (CDAI)≤ 10.
Percentage of remission (CDAI) at week 12 | At week 12
  Remission is defined as crohn's disease activity index (CDAI)≤ 2.8.

SECONDARY OUTCOMES:
Percentage of low disease activity (DAS28-CRP) at week 12 | March 1, 2021
  Low disease activity is defined as DAS28-CRP score ≥ 2.6 but ≤ 3.2
Patient disease activity assessment (VAS) at week 12 | at week 12
  based on a scale of 0=no disease to 10=severe disease
Patient Pain Global assessment (VAS) at week 12 | at week 12
  based on a scale of 0=no disease to 10=severe disease
Function evaluation at week 12 | at week 12
  Health Assessment Questionnaire Disability Index (HAQ-DI) for function evaluation
Medication possession rate (MPR) at week 12 | at week 12
Medication possession rate (MPR) at week 24 | at week 24
Medication possession rate (MPR) at week 48 | at week 48

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China